CLINICAL TRIAL: NCT00487513
Title: Procurement of Follicular B Cell Lymphoma Cells From Blood, Tissue or Malignant Effusion for the Purpose of Possible Use in Future Clinical Trials: A Minimal Risk Protocol
Brief Title: Procurement of Follicular B Cell Lymphoma Cells for the Purpose of Possible Use in Future Clinical Trials
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Eric Jacobsen, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 06-276
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Follicular B Cell lymphoma; vaccination
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Lymph node biopsy Drainage of an effusion Bone marrow biopsy
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Procurement of Follicular B Cell Lymphoma Cells — Participants will undergo the following procedure(s) that are appropriate for collecting their tissue: Blood collection, lymph node biopsy, drainage of an effusion, or bone marrow biopsy

SUMMARY:
In order to learn more about follicular lymphoma and anti-cancer vaccines, we are collecting samples from people with this diagnosis. We then hope to make a vaccine from this tissue to help the immune system destroy cancer cells. We plan on keeping samples in the tissue bank indefinitely.

DETAILED DESCRIPTION:
- The following tests and procedures will be performed: Approximately 50cc of peripheral blood will be drawn and stored in the tissue bank; patients who have follicular lymphoma cells circulating in the blood will have about 40cc's of blood drawn and stored for processing; patients undergoing a lymph node biopsy will have samples of the biopsy stored; patients having fluid drained from the abdomen or from around the lung will have some of their fluid saved to cell collection and processing; patients undergoing a bone marrow biopsy will have some of the sample stored for cell collection and processing.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed, refractory or de novo histologically confirmed follicular B-cell lymphoma with accessible lymph nodes, tumor mass or malignant effusion or peripheral blood
* 35 years of age or older

Exclusion Criteria:

* Uncontrolled active infection
* HIV or viral Hepatitis infection
* Other current malignancies except any in situ cancer or basal or squamous cell carcinoma of the skin
* Autoimmune cytopenias

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are selected because they have Non-Hodgkin's lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Tissue collection for vaccine generation | 2 years
  Collect eligible patient samples that potentially could be used to prepare autologous cell vaccines and possibly prepare autologous tumor cell injection for vaccine induced delayed-type hypersensitiviy evaluation for the companion treatment protocol. There will be no analysis performed on this protocol, the analysis will occur on a companion vaccination protocol. Patients will be consented to this protocol separately.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States